CLINICAL TRIAL: NCT04549727
Title: Development and Use of a Tissue and Human Enteroid Biorepository to Study the Pathophysiology of Neonatal Necrotizing Enterocolitis
Brief Title: Development and Use of a Tissue and Human Enteroid Biorepository to Study the Pathophysiology of NEC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BIENTERNIP
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Enterocolitis, Necrotizing; Prematurity; Gastrointestinal Disease
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infants with surgical NEC: Infants who undergo surgery for NEC disease
  Interventions: Other: Organoids creation
- Infants with GI surgical diseases other than NEC: Infants who undergo surgery for other GI diseases than NEC
  Interventions: Other: Organoids creation

INTERVENTIONS:
Other: Organoids creation — Organoids are created from discarded tissue

SUMMARY:
Despite a greater understanding of NEC physiopathology, modest progress has been done in terms of intervention and prevention of the disease over the past three decades, being the mortality rate unchanged.

Investigators intend to leverage our knowledge and technical expertise developed with fetal enteroids to further investigate the processes leading to NEC by deriving and performing functional studies on human intestinal enteroids generated from intestinal resection for therapeutic reasons in NEC and non-NEC patients

1. Generate a tissue biorepository composed of: enteroids and other lamina propria cells
2. Comparative studies of the gene expression profile of tissue, epithelial enteroids and underlying lamina propria of NEC, non-NEC, hypoxic and non-hypoxic infants
3. In vitro functional studies for the evaluation of critical factors in NEC pathophysiology
4. In vitro functional studies to identify the activation of processes leading to intestinal epithelium necroptosis and/or apoptosis in bacteria challenged and hypoxic conditions
5. Correlative studies of the impact of perinatal variables on the intestinal barrier functionality at baseline and challenged with pathogens
6. In vitro comparison of the intestinal barrier functionality in infants complicated by condition of prenatal hypoxia versus non hypoxic infants
7. Validation the NEC enteroids as an in vitro model for the identification of treatments and prevention of NEC

ELIGIBILITY:
Inclusion Criteria:

* Infants, with a postconceptional age below 44 weeks of gestation, undergoing a clinically indicated intervention of partial intestinal resection while hospitalized at the NICU of the Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico.

Exclusion Criteria:

* Infants presenting a devastating damage of the intestine

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Investigators will use surgically-resected intestinal samples from NEC patients and gestational age-matched non-NEC surgical controls with intestinal resection for other reasons than NEC to conduct various analysis. For comparative studies, Investigators aim to grow enteroids from intestinal tissues freshly collected from preterm and term babies with an age limit of 44 weeks of postmenstrual age (PMA).
  Group 1: intestinal samples from small and/or large bowel in NEC preterm and term babies.
  Group 2 (Control group): Age- and intestinal area-matched (small and/or large bowel) No NEC babies, which have surgical resection for other reason than NEC
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-02-17 (Estimated); Study Completion 2022-02-17 (Estimated)

PRIMARY OUTCOMES:
Comparative studies of gene expression | 2 years
  assess the gene expression profile of tissue, epithelial enteroids and underlying lamina propria derived from NEC, non-NEC (further classified as hypoxic and non-hypoxic infants).
  NB: the unit of analysis will be the organoids derived from patients' tissues Investigators expect to be able to derive 1 cell line per patient, and the number of derived organoids will depend from the viability of individual cell lines.
functional studies barrier functionality | 2 years
  evaluation of barrier functionality at the baseline and in enteroids-derived monolayers challenged with pathogens, dead bacteria (as postbiotics), LPS, pharmacological agents, enteral nutrients and to evaluate innate immune response and barrier functionality as previously investigated in fetal enteroids and the contribution of myofibroblast, immune and ENS to the immune response
functional studies on cellular death | 2 years
  studies to identify the activation of processes leading to intestinal epithelium necroptosis and/or apoptosis in bacteria challenged and hypoxic conditions
Correlative studies of the impact of perinatal variables | 2 years
  Assess how the perinatal features (expression of the neonatal phenotype, as IUGR, chorionamnionitis, perinatal hypoxia) on the intestinal barrier functionality at baseline and challenged with pathogens
compare the intestinal barrier functionality in pathological conditions | 2 years
  comparison of the intestinal barrier functionality in infants complicated by condition of prenatal hypoxia versus non hypoxic infants
Validation of the enteroid NEC model | 2 years
  Validate the NEC enteroids as an in vitro model for the identification of treatments and prevention of NEC.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Roggero, MD PHD, Principal Investigator — University of Milan Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico

IPD SHARING:
Plan to Share IPD: Undecided